CLINICAL TRIAL: NCT06788561
Title: Effect of Non-invasive Transcutaneous Vagus Nerve Stimulation for Pain Control After Cesarean Delivery - a Randomised Controlled Trial
Brief Title: Effect of Transcutaneous Vagus Nerve Stimulation for Pain Control After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TREC2024-KY089.R1
Record Dates: First submitted 2024-12-19; First posted 2025-01-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain, Acute
Keywords: Transcutaneous auricular vagus nerve stimulation (taVNS); Auricular acupoint; Cesarean section; Postoperative pain; Inflammatory response
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcutaneous auricular vagus nerve stimulation (taVNS) (Experimental): Bilateral auricle area is selected, where the branches of the vagus nerve are abundantly distributed. The use of an SDZ-IIB electronic acupuncture therapy device and specially designed ear clips to stimulate both sides for 30 minutes each session. The stimulation parameters are set to sparse dense wave, with a frequency of 4 Hz/20 Hz, and the intensity is adjusted based on the patient's tolerance, gradually increasing from 0 to the highest point the patient can tolerate. A total of two stimulations are administered, the first immediately after the baby is delivered, and the second is 23.5 hours postoperative.
  Interventions: Device: Transauricular Nerve Stimulation
- Sham transcutaneous auricular vagus nerve stimulation (s-taVNS) (Sham Comparator): Bilateral auricular areas are selected, where the branches of the vagus nerve are abundantly distributed. An SDZ-IIB electronic acupuncture therapy device and specially designed ear clips are used to stimulate both sides. The stimulation parameters are set to sparse dense waves, with a frequency of 4 Hz/20 Hz, and the intensity is adjusted based on the patient's tolerance, gradually increasing from 0 to the highest level the patient can endure, then the device is then turned off, electric current stimulation is applied for approximately 10 seconds. The process of attaching the clip to the earlasts for 30 minutes. A total of two stimulations are administered, the first immediately after the baby is delivered, and the second 23.5 hours postoperatively.
  Interventions: Device: s-taVNS

INTERVENTIONS:
Device: Transauricular Nerve Stimulation — Hua Tuo brand SDZ-IIB electronic acupuncture therapy device and specially designed ear clips.
  Arms: Transcutaneous auricular vagus nerve stimulation (taVNS)
Device: s-taVNS — Hua Tuo brand SDZ-IIB electronic acupuncture therapy device and specially designed ear clips.
  Arms: Sham transcutaneous auricular vagus nerve stimulation (s-taVNS)

SUMMARY:
This study investigates whether non-invasive transcutaneous auricular vagus nerve stimulation can alleviate postoperative pain in patients after cesarean section, and explores its possible mechanisms of action through an exploratory study.

DETAILED DESCRIPTION:
Post-cesarean section pain, if improperly managed, may affect the prognosis of the mother and the health of the infant. There is an urgent need to explore safer, more effective, and more direct non-pharmacological, non-invasive adjunctive interventions to alleviate the pain associated with cesarean section. Non-invasive transcutaneous auricular vagus nerve stimulation is a green neuromodulatory measure that has shown significant improvement in various types of pain and holds great potential for relieving perioperative pain. This study aims to investigate whether non-invasive transcutaneous auricular vagus nerve stimulation can alleviate postoperative pain in patients after cesarean section and to explore the possible mechanisms by which it exerts its effects, through a prospective randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are classified as American Society of Anesthesiologists (ASA) physical status I to III.
2. Scheduled for elective cesarean delivery under spinal anesthesia.
3. Patients are aged between 19 to 45 years old.
4. Patients have provided written informed consent.

Exclusion Criteria:

1. Local skin infection occurs in the auricular area during transcutaneous auricular vagus nerve stimulation.
2. Cases where spinal anesthesia fails and general anesthesia is required.
3. Patients with conditions such as recurrent alcohol abuse, fever, convulsions, or cardiopulmonary failure.
4. Patients who have used opioid medications at least 6 months prior to surgery.
5. Patients who are unable to understand the consent form and study questionnaire, including those with cognitive impairments.
6. Patients with a history of psychiatric illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS-11) pain score during movement | 24 hours postoperatively
  Numeric Rating Scale (NRS-11), this scale is a validated tool for measuring pain intensity, with scores ranging from 0 (no pain) to 10 (the most severe pain imaginable).The higher the score, the more severe the pain.

SECONDARY OUTCOMES:
the proportion of patients with NRS pain score > 6 | 24 hours postoperatively
  Assess the proportion of severe pain by calculating the ratio of NRS pain scores that are greater than 6.
Epinephrine | 48 hours postoperatively
  Serum Epinephrine concentration.
C-reactive protein (CRP) | 48 hours postoperatively
  Serum CRP concentration.
NFκB | 48 hours postoperatively
  Serum NFκB concentration.
aEP | 48 hours postoperatively
  Serum aEP concentration
Postoperative adverse reactions | From date of randomization until the date of discharge, assessed up to 7 days
  Explore whether taVNS intervention increases postoperative adverse reactions, including dizziness, bloating, itching and so on.
Postoperative severe complications | From date of randomization until the date of discharge, assessed up to 7 days
  Postoperative severe complications, including pulmonary complications, liver function abnormalities, heart function abnormalities, kidney function abnormalities, and SIRS (Systemic Inflammatory Response Syndrome).

CONTACTS AND LOCATIONS:
Overall Officials: Guyan Wang, Study Director — Beijing Tongren Hospital
Locations (1):
- Beijing tongren Hospital, Capital Medical University, Beijing, China